CLINICAL TRIAL: NCT01378052
Title: Level of DNA Methylation in People With Urothelial Carcinoma
Brief Title: DNA Methylation and Urothelial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Chao-Hsiang Chang, Department of Urology
Other Study IDs: DMR100-IRB-092
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- urothelial carcinoma pateints
- healthy controls: Age and gender matched control subjects with no evidence of UC or any other malignancy were accrued from the hospital, recruiting people receiving adult health examinations at China Medical University Hospital.

SUMMARY:
Many studies previously showed the significant association between urinary arsenic profiles and urothelial carcinoma (UC) risk and observed the increased UC risk in people with lower plasma folate and higher homocysteine than those with higher plasma folate and lower homocysteine. The investigators would expect to explore the interactions among global DNA methylation, one-carbon metabolic pathway factors, urinary arsenic profiles and UC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urothelial carcinoma
* The voluntary of participating the study

Exclusion Criteria:

* Age smaller than 20 years
* Pregnant women
* Not willing to participate the study because of their personal reasons

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a hospital-based case-control study. Patients with urothelial carcinoma are recruited by pathological verification of UC was done by routine urological practice including endoscopic biopsy or surgical resection of urinary tract tumors followed by histopathological examination by board-certified pathologists. Healthy controls without evidence of UC or any other malignancy were recruited including those receiving adult health examinations at China Medical University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
urothelial carcinoma | one year
  Pathological verification of UC was done by routine urological practice including endoscopic biopsy or surgical resection of urinary tract tumors followed by histopathological examination by board-certified pathologists.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Jung Chung, PhD, Principal Investigator — Department of Health risk Management, China Medical University
Locations (1):
- Department of Urology, China Medical University Hospital, Taichung, 404, Taiwan